CLINICAL TRIAL: NCT04861714
Title: Evaluation of Regeneten Augmentation for Subscapularis Healing After Total Shoulder Arthroplasty (RESTOR)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Cvetanovich, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019H0419
Record Dates: First submitted 2021-02-11; First posted 2021-04-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Regeneten (Active Comparator): Standard subscapularis repair with Regeneten augmentation group
  Interventions: Device: Regeneten
- Standard repair (Other): Standard subscapularis repair
  Interventions: Procedure: Standard repair

INTERVENTIONS:
Device: Regeneten — Augmentation of standard subscapularis repair with regeneten patch
  Arms: Regeneten
Procedure: Standard repair — Standard subscapularis repair
  Arms: Standard repair

SUMMARY:
The purpose of this study is to evaluate whether augmentation of subscapularis repair with the Regeneten implant after anatomic total shoulder arthroplasty (TSA) can improve rates of subscapularis healing and improve clinical outcomes.

DETAILED DESCRIPTION:
Subscapularis management is an area of controversy in the literature for total shoulder arthroplasty (TSA). Regeneten has been suggested as a bioinductive implant to aid in rotator cuff healing. We hypothesize that applying this technology could aid in obtaining higher rates of subscapularis healing for TSA when utilizing SP or ST, which in turn could lead to improved outcomes.The 50 randomized subjects will be randomized at a 1:1 ratio into the standard subscapularis repair group or the standard repair with Regeneten augmentation group. Subjects will be blinded to their treatment assignment until they complete all study visits. Upon withdraw from the study, termination from the study, or new or recurrent symptoms requiring a subsequent surgical procedure, the blinded assignment will be revealed to the subject. Subjects will be assessed pre-operatively and return post-operatively at Week 2, Weeks 6, Month 3, Month 6, and Year 1. The primary outcome will evaluate subscapularis repair integrity and healing at one year post-op.

ELIGIBILITY:
Inclusion Criteria:

1. Patients healthy enough to undergo primary anatomic TSA
2. Being treated with subscapularis tenotomy or subscapularis peel.
3. Age 50 or above
4. Intact rotator cuff including subscapularis as determined by preoperative examination and imaging (typically preoperative CT, MRI if indicated or available).

Exclusion Criteria:

1. Revision arthroplasty
2. Reverse arthroplasty
3. Requiring a lesser tuberosity osteotomy
4. Intraoperative identification of rotator cuff tear requiring repair
5. Object to using cow derived material
6. Prior index shoulder surgery requiring treatment to the subscapularis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Subscapularis repair integrity assessed by lift-off test using dynamometry. | 12 months post-op
  Pounds (lbs) of force that the subject can produce during the lift off test will be recorded.

SECONDARY OUTCOMES:
Forward elevation active range of motion as assessed by treating physician | 6 weeks
  The amount of forward elevation range of motion will be reported in degrees from 0-180.
Forward elevation active range of motion as assessed by treating physician | 3 months
  The amount of forward elevation range of motion will be reported in degrees from 0-180.
Forward elevation active range of motion as assessed by treating physician | 6 months
  The amount of forward elevation range of motion will be reported in degrees from 0-180.
Forward elevation active range of motion as assessed by treating physician | 12 months
  The amount of forward elevation range of motion will be reported in degrees from 0-180.
Abduction active range of motion as assessed by treating physician | 6 weeks
  The amount of abduction range of motion will be reported in degrees from 0-180.
Abduction active range of motion as assessed by treating physician | 3 months
  The amount of abduction range of motion will be reported in degrees from 0-180.
Abduction active range of motion as assessed by treating physician | 6 months
  The amount of abduction range of motion will be reported in degrees from 0-180.
Abduction active range of motion as assessed by treating physician | 12 months
  The amount of abduction range of motion will be reported in degrees from 0-180.
External rotation active range of motion as assessed by treating physician | 6 weeks
  The amount of external rotation range of motion will be reported in degrees from 0-180.
External rotation active range of motion as assessed by treating physician | 3 months
  The amount of external rotation range of motion will be reported in degrees from 0-180.
External rotation active range of motion as assessed by treating physician | 6 months
  The amount of external rotation range of motion will be reported in degrees from 0-180.
External rotation active range of motion as assessed by treating physician | 12 months
  The amount of external rotation range of motion will be reported in degrees from 0-180.
Internal rotation active range of motion as assessed by treating physician | 6 weeks
  The amount of internal rotation range of motion will be reported in vertebrae level the thumb reaches from 0, 0°; 1, hip; 2, buttocks; 3, sacrum; 4, L4-L5; 5, L1-L3; 6, T8-T12; 7, T7 or higher.
Internal rotation active range of motion as assessed by treating physician | 3 months
  The amount of internal rotation range of motion will be reported in vertebrae level the thumb reaches from 0, 0°; 1, hip; 2, buttocks; 3, sacrum; 4, L4-L5; 5, L1-L3; 6, T8-T12; 7, T7 or higher.
Internal rotation active range of motion as assessed by treating physician | 6 months
  The amount of internal rotation range of motion will be reported in vertebrae level the thumb reaches from 0, 0°; 1, hip; 2, buttocks; 3, sacrum; 4, L4-L5; 5, L1-L3; 6, T8-T12; 7, T7 or higher.
Internal rotation active range of motion as assessed by treating physician | 12 months
  The amount of internal rotation range of motion will be reported in vertebrae level the thumb reaches from 0, 0°; 1, hip; 2, buttocks; 3, sacrum; 4, L4-L5; 5, L1-L3; 6, T8-T12; 7, T7 or higher.
Patient reported clinical outcome scores on the American Shoulder and Elbow Surgeon Evaluation (ASES) | 6 weeks
  The American Shoulder and Elbow Surgeons (ASES) score is composed of a patient-reported portion and a physician assessment.The ASES tool includes a patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
Patient reported clinical outcome scores on the American Shoulder and Elbow Surgeon Evaluation (ASES) | 3 months
  The American Shoulder and Elbow Surgeons (ASES) score is composed of a patient-reported portion and a physician assessment.The ASES tool includes a patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
Patient reported clinical outcome scores on the American Shoulder and Elbow Surgeon Evaluation (ASES) | 6 months
  The American Shoulder and Elbow Surgeons (ASES) score is composed of a patient-reported portion and a physician assessment.The ASES tool includes a patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
Patient reported clinical outcome scores- American Shoulder and Elbow Surgeon Evaluation (ASES) | 12 months
  The American Shoulder and Elbow Surgeons (ASES) score is composed of a patient-reported portion and a physician assessment.The ASES tool includes a patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
Patient reported clinical outcome scores- Visual Analog Scale (VAS) | 6 weeks
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. Score ranges from 0-100mm where 0mm= no pain and 100mm=extreme pain.
Patient reported clinical outcome scores- Visual Analog Scale (VAS) | 3 months
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. Score ranges from 0-100mm where 0mm= no pain and 100mm=extreme pain.
Patient reported clinical outcome scores- Visual Analog Scale (VAS) | 6 months
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. Score ranges from 0-100mm where 0mm= no pain and 100mm=extreme pain.
Patient reported clinical outcome scores- Visual Analog Scale (VAS) | 12 months
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. Score ranges from 0-100mm where 0mm= no pain and 100mm=extreme pain.
Patient reported clinical outcome scores- Simple shoulder test (SST) | 6 weeks
  The simple shoulder test is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. Answers of 'yes' receive a score of 1 and answers of 'no' receive a score of 0. Scores range from 0-12 where 0=no function and 12=full function.
Patient reported clinical outcome scores- Simple shoulder test (SST) | 3 months
  The simple shoulder test is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. Answers of 'yes' receive a score of 1 and answers of 'no' receive a score of 0. Scores range from 0-12 where 0=no function and 12=full function.
Patient reported clinical outcome scores- Simple shoulder test (SST) | 6 months
  The simple shoulder test is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. Answers of 'yes' receive a score of 1 and answers of 'no' receive a score of 0. Scores range from 0-12 where 0=no function and 12=full function.
Patient reported clinical outcome scores- Simple shoulder test (SST) | 12 months
  The simple shoulder test is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. Answers of 'yes' receive a score of 1 and answers of 'no' receive a score of 0. Scores range from 0-12 where 0=no function and 12=full function.
Patient reported clinical outcome scores- Simple shoulder value (SST) | 6 weeks
  The simple shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.
Patient reported clinical outcome scores- Simple shoulder value (SST) | 3 months
  The simple shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.
Patient reported clinical outcome scores- Simple shoulder value (SST) | 6 months
  The simple shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.
Patient reported clinical outcome scores- Simple shoulder value (SST) | 12 months
  The simple shoulder value is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cvetanovich, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Sports Medicine Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.